CLINICAL TRIAL: NCT03476187
Title: Benefits of µCor in Ambulatory Decompensated Heart Failure
Acronym: BMADHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 90D0182
Record Dates: First submitted 2018-02-19; First posted 2018-03-23 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- µCor wearers (Experimental): Wear the µCor device
  Interventions: Device: µCor

INTERVENTIONS:
Device: µCor — Monitor with µCor

SUMMARY:
Subjects meeting the inclusion/exclusion criteria will wear the µCor for at least 90 days. During the study, clinic follow up will occur every 30 days. For all subjects, each scheduled clinic visit will include assessment of cardiac symptoms and any relevant clinically actionable events. The subject will be given a daily diary to track symptoms, unplanned hospital visits, medication changes, and all other heart failure related clinical events. Weekly phone calls to the subject will be given throughout the duration of the study to remind the patient to use the subject diary and to collect and record heart failure related clinical events. Subjects will be contacted six months and one year from initial enrollment to assess the vital status of the subject, any heart failure related clinical events since the end of µCor wear, and any health care utilization since the end of µCor wear.

DETAILED DESCRIPTION:
Subjects meeting the inclusion/exclusion criteria will wear µCor for 90 days from the day of fitting. 500 total patients will be enrolled. There will be an interim analysis when the 200th subject has finished the study in the study to assess for distribution of patients with reduced and preserved LVEF.

Subjects will be fitted with µCor during hospital discharge or within a clinic visit that has occurred within 10 days of a heart failure related hospitalization. The µCor fitting will mark day 0 of the study. An LVEF measurement will be recorded during enrollment or within 30 days post enrollment if an LVEF measurement has not been recorded within 30 days prior to enrollment. An investigator assessment will be performed during all clinic visits. The assessment template is shown in Appendix A.

Subjects will be given a diary at enrollment that will ask them to rate their degree of specific symptoms of heart failure such as shortness of breath and fatigue as well as mark any heart failure related clinical events or medication changes that have occurred since the last entry.

Study follow up visits will occur at day 30, day 60, and day 90. During follow up visits the subjects will be asked about any heart failure related clinical events or change in symptoms that have occurred since the last follow up. The subject will receive a study based weekly phone call asking the subject about any recent heart failure related clinical events or change in heart failure symptoms. During the weekly phone call the subject will be reminded to fill out the daily diary. No phone calls will be given on the week where there is a study follow up visit. There will be 9 total phone calls.

During the Day 90 visit, the subject will be given the option to continue wearing the µCor for an additional 90 days. Furthermore, if the subject experienced a heart failure related clinical event within the initial 90 days of wear, the subject will be given the option of wearing the µCor for 30 days following the heart failure event. .If the subject chooses additional wear time, weekly phone calls and monthly visits will be structured identical to that of the main study period. The µCor will be returned at end of use.

There will be a follow up at six months and one year post enrollment to document mortality data, heart failure related clinical events, and health care utilization data.

ELIGIBILITY:
Inclusion Criteria:

* Subjects either hospitalized for decompensated systolic, diastolic, or combined heart failure or subjects presenting at an outpatient clinic with a history of hospital discharge for decompensated systolic, diastolic, or combined heart failure within the previous 10 days.
* All subjects must be 21 years of age or older on the day of screening.

Exclusion Criteria:

* Subjects who are wearing the wearable cardioverter defibrillator (WCD)
* Subjects not expected to survive one year from enrollment from non-cardiac disease.
* Subjects with skin allergy or sensitivity to medical adhesives.
* Subjects anticipated to start dialysis within 90 days.
* Subjects currently implanted with an S-ICD system.
* Subjects whose primary diagnosis on hospital admission was Acute Coronary Syndrome (ACS) STEMI/NSTEMI rather than heart failure exacerbation.
* Subjects who are unable to participate in all follow up visits.
* Subjects participating in any other research at time of enrollment.
* Subjects currently implanted with an LVAD.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Szymkiewicz, MD, Study Director — Zoll Medical Corporation
Locations (61):
- United States (57):
  - Mobile Heart Specialists, PC, Mobile, Alabama
  - University Hospital, Mobile, Alabama
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Cardiovascular Innovation and Research Center, Inc., Long Beach, California
  - Los Alamitos Cardiovascular, Los Alamitos, California
  - Nova Clinical Research LLC, Bradenton, Florida
  - South Palm Cardiovascular Research Institute, Delray Beach, Florida
  - Holy Cross Medical Group, Fort Lauderdale, Florida
  - The Cardiac and Vascular Institute Research Foundation, Gainesville, Florida
  - Baptist Heart Specialists, Jacksonville, Florida
  - The Heart Institute at Largo, Largo, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Cardiovascular Institute of Central Florida, Ocala, Florida
  - Northside Hospital, St. Petersburg, Florida
  - University of South Florida Dept of Cardiovascular Sciences, Tampa, Florida
  - Cardiology Practice Tampa, Tampa, Florida
  - Cardiovascular Consultants of South Georgia, Thomasville, Georgia
  - Fox Valley Clinical Research Center, Aurora, Illinois
  - The Loretto Hospital, Chicago, Illinois
  - Chicago Medical Research LLC, Hazel Crest, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Unity Point Health Cardiovascular Services, Peoria, Illinois
  - DuPage Medical Group, Winfield, Illinois
  - Grace Research LLC, Bossier City, Louisiana
  - Clinical Trials of America, LLC, Monroe, Louisiana
  - Clinical Trials of America, LLC, West Monroe, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cardiology Institute of Michigan, Flint, Michigan
  - Hennepen Healthcare Research Institute, Minneapolis, Minnesota
  - Nebraska Heart Institute, Grand Island, Nebraska
  - Nebraska Heart Institute, Lincoln, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - New Jersey Heart, Linden, New Jersey
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Trinity Medical WNY, Buffalo, New York
  - SJH Cardiology Associates, Liverpool, New York
  - University of Rochester Medical Center, Rochester, New York
  - East Carolina Heart Institute, Greenville, North Carolina
  - NC Heart & Vascular Research, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - OUHSC, Oklahoma City, Oklahoma
  - UMPC Hamot, Erie, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - The Guthrie Clinic, Sayre, Pennsylvania
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - Palmetto Health Advanced Heart Health Center, Columbia, South Carolina
  - The Jackson Clinic, PA, Jackson, Tennessee
  - PharmaTex Research, Amarillo, Texas
  - JPS Health Network, Fort Worth, Texas
  - Texas Cardiovascular Institute, Fort Worth, Texas
  - Northwest Houston Cardiology, Houston, Texas
  - CardioVogage, McKinney, Texas
  - Texas Institute of Cardiology, McKinney, Texas
  - Riverside Hospital Inc., Newport News, Virginia
  - Chippenham Hospital, Richmond, Virginia
  - Henrico Doctors Hospital, Richmond, Virginia
  - Marshall Cardiology, Huntington, West Virginia
- Universitätsklinik für Innere Medizin II, Abteilung für Kardiologie, Vienna, Austria
- Germany (3):
  - St. Vinzenz-Hospital; Akademisches Lehrkrankenhaus der Universität zu Köln, Innere Medizin III, Cologne
  - Herzzentrum Leipzig GmbH, Leipzig
  - Klinikum rechts der Isar - Technische Universität München, Klinik und Poliklinik für Innere Medizin I, Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boehmer JP, Cremer S, Abo-Auda WS, Stokes DR, Hadi A, McCann PJ, Burch AE, Bonderman D. Impact of a Novel Wearable Sensor on Heart Failure Rehospitalization: An Open-Label Concurrent-Control Clinical Trial. JACC Heart Fail. 2024 Dec;12(12):2011-2022. doi: 10.1016/j.jchf.2024.07.022. Epub 2024 Oct 9. PMID 39387771

RESULTS

PARTICIPANT FLOW:
Groups:
- µCor Wearers: Subjects wearing the µCor device
Period: Overall Study
Arm/Group | µCor Wearers
Started | 257
Completed | 245
Not Completed | 12
Not completed — Protocol Violation | 7
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | µCor Wearers
Number analyzed (Participants) | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 144
Race/Ethnicity, Customized [Number; unit: participants]
  Ethnicity : Caucasian | 154
  Ethnicity : Black or African American | 62
  Ethnicity : Hispanic or Latin | 16
  Ethnicity : Other | 5
  Ethnicity : American Indian or Alaskan Native | 2
  Ethnicity : Asian | 1
  Ethnicity : Don't Know / No Response | 1
  Ethnicity: Multiple Ethnicities | 4
Region of Enrollment [Number; unit: participants]
  Austria | 13
  United States | 221
  Germany | 11
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.6 (10.4)
Blood Pressure (systolic) [Mean (Standard Deviation); unit: mmHg] | 122.1 (19.3)
Blood Pressure (diastolic) [Mean (Standard Deviation); unit: mmHg] | 71.5 (12.2)
Respiration Rate [Mean (Standard Deviation); unit: breaths per min] | 18.1 (2.8)
Heart Rate [Mean (Standard Deviation); unit: beats per min] | 77 (14.5)
Years from Heart Failure Diagnosis [Mean (Standard Deviation); unit: years] | 4.2 (6.2)
Left Ventricular Ejection Fraction (Minimum) [Mean (Standard Deviation); unit: % of blood ejected from left ventricle] | 38.7 (17.4)
Left Ventricular Ejection Fraction (Maximum) [Mean (Standard Deviation); unit: % of blood ejected from left ventricle] | 42.1 (17.2)
Cardiac Device History [Count of Participants; unit: Participants]
  History of Pacemaker: Yes | 54
  History of Pacemaker: No | 191
  History of Pacemaker: Unknown | 0
  Pacemaker Active: Yes | 50
  Pacemaker Active: No | 4
  Pacemaker Active: Unknown | 191
  History of ICD: Yes | 72
  History of ICD: No | 173
  History of ICD: Unknown | 0
  ICD Active: Yes | 67
  ICD Active: No | 5
  ICD Active: Unknown | 173
  Current Heart Failure Monitoring System: Yes | 8
  Current Heart Failure Monitoring System: No | 237
  Current Heart Failure Monitoring System: Unknown | 0
Heart Failure Etiology [Count of Participants; unit: Participants]
  Ischemic | 93
  Non-ischemic | 136
  Mixed | 16
Medical History [Count of Participants; unit: Participants]
  History of Hypertension: Yes | 222
  History of Hypertension: No | 22
  History of Hypertension: Unknown | 1
  History of Diabetes: Yes | 142
  History of Diabetes: No | 103
  History of Diabetes: Unknown | 0
  History of COPD: Yes | 95
  History of COPD: No | 146
  History of COPD: Unknown | 4
  History of Transient Ischemic Attack: Yes | 52
  History of Transient Ischemic Attack: No | 189
  History of Transient Ischemic Attack: Unknown | 4
  History of Chronic Kidney Disease: Yes | 107
  History of Chronic Kidney Disease: No | 134
  History of Chronic Kidney Disease: Unknown | 4
  History of Angina: Yes | 75
  History of Angina: No | 161
  History of Angina: Unknown | 9
  History of Syncope: Yes | 43
  History of Syncope: No | 192
  History of Syncope: Unknown | 10
  History of Sudden Cardiac Arrest: Yes | 8
  History of Sudden Cardiac Arrest: No | 234
  History of Sudden Cardiac Arrest: Unknown | 3
  History of Arrhythmia: Yes | 155
  History of Arrhythmia: No | 81
  History of Arrhythmia: Unknown | 9
  History of Myocardial Infarction: Yes | 78
  History of Myocardial Infarction: No | 155
  History of Myocardial Infarction: Unknown | 12
  History of Coronary Artery Bypass Graft (CABG): Yes | 49
  History of Coronary Artery Bypass Graft (CABG): No | 194
  History of Coronary Artery Bypass Graft (CABG): Unknown | 2
  History of Percutaneous Coronary Intervention (PCI): Yes | 74
  History of Percutaneous Coronary Intervention (PCI): No | 165
  History of Percutaneous Coronary Intervention (PCI): Unknown | 6
New York Heart Classification [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Functional Classification places patients in 1 of 4 categories based on limitations of physical activity. The healthcare practitioner assigns the patient.
  I= No limitation of physical activity. II= Slight limitation of physical activity. III= Marked limitation of physical activity. IV= Symptoms of heart failure at rest- Any physical activity causes further discomfort.
  Participants
    Class I | 3
    Class II | 69
    Class III | 122
    Class IV | 9
    Not documented | 42

OUTCOME MEASURES:

1. Primary Outcome: Correlation of μCor Readings to Heart Failure Related Clinical Events
Description: HF Event: a hospitalization primarily due to heart failure within 90 days. Time window: The 7 days prior to the 1st heart failure hospitalization, or the final 7 days of device wear if no HF event occurred.
Time Frame: 3 months
Population: The median of each device value was calculated for each subject within their time window. ROC analysis was performed. Data are presented assuming that the device reading in subjects without HF events < that of subjects with HF events.
Measure: Number; unit: participants
Arm/Group | µCor Wearers
Number analyzed (Participants) | 245
participants
  Valid device data within time window : HF Event | 34
  Valid device data within time window : No HF Event | 173
  No valid device data within time window : HF Event | 16
  No valid device data within time window : No HF Event | 22

2. Primary Outcome: Correlation of µCor Readings to Heart Failure Related Clinical Events
Description: Definitions:
  Daytime: 7:00 AM - 12:00 AM Nighttime: 12:00 AM - 7:00 AM
  For each day on which the subject wore the device, the following values were calculated:
  Daytime activity: The proportion of minutes while wearing the device that the subject spent active (unitless).
  Nighttime heart rate: The median heart rate while wearing the device during the night (beats/min)
  Thoracic fluid index: The median proportion of ratio of radiofrequency-measured lung fluid readings compared to the subject's baseline (unitless).
  Nighttime posture: The median pitch angle while wearing the device during the night (degrees, where 0 is the horizontal).
  Nighttime respiration: The median respiration rate while wearing the device during the night (breaths/min)
  HF event: a hospitalization primarily due to heart failure
Time Frame: 3 months
Population: The median was calculated for the 7 days prior to the 1st hospitalization; the median was calculated for the final 7 days of device wear. ROC analysis was performed. Data are presented assuming that the device reading in subjects without events is less than that of subjects with events. Unit of measure: probability that a randomly chosen subject with a HF event has a greater device value than a randomly chosen subject without a HF event.
Measure: Median (95% Confidence Interval); unit: Probability
Arm/Group | µCor Wearers
Number analyzed (Participants) | 245
Probability
  Daytime Activity | 0.35 [0.26 to 0.45]
  Nighttime Heart Rate | 0.59 [0.48 to 0.70]
  Thoracic Fluid Index | 0.59 [0.49 to 0.68]
  Nighttime Posture | 0.59 [0.49 to 0.70]
  Nighttime Respiration | 0.59 [0.48 to 0.70]

3. Secondary Outcome: Establishment of Rate of Occurrence of VT/VF Episodes and Arrhythmic Death in Subjects
Description: Rate of occurrence of VT/VF episodes at the time of enrollment in the study and rate of occurrence of arrhythmic death in subjects at 90 days and 1 year.
Time Frame: Baseline, 90 days, 1 YR
Population: Rate of occurrence of VT/VF episodes at the time of enrollment in the study and rate of occurrence of arrhythmic death at 90 days and 1 year
Measure: Number; unit: participants
Arm/Group | µCor Wearers
Number analyzed (Participants) | 245
participants
  VT at baseline | 10
  VF at baseline | 3
  VT (non-sustained) at baseline | 12
  Arrhythmic death at 1 year | 2
  Arrhythmic death at 90 days | 1

4. Secondary Outcome: Correlation Between μCor Measurements and Subject Reported Symptoms - Area Under Curve
Description: During office visits at months 1, 2, and 3, subjects reported their degrees of dyspnea, orthopnea, and fatigue on the following scale: [none, seldom, frequent, continuous]. Each day that the subject wore the device, a daily median was calculated for the following measures: [thoracic fluid index (TFI), nighttime heart rate (HR), nighttime respiration rate (RR)]. Nighttime was defined as 12:00 AM - 7:00 AM.
Time Frame: 3 months
Population: The median of the daily medians for each device measure was calculated for the 7 days preceding each office visit. To assess whether reports of severe [frequent or continuous] symptoms were associated with greater device measures than reports of mild symptoms [none or seldom], receiver operating characteristic (ROC) analysis was performed. Unit of measure: probability a randomly chosen subject with severe symptoms has a greater device value than a randomly chosen subject with mild symptoms.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | µCor Wearers
Number analyzed (Participants) | 245
Probability
  Dyspnea - TFI | 0.56 [0.49 to 0.62]
  Dyspnea - HR | 0.53 [0.46 to 0.60]
  Dyspnea - RR | 0.47 [0.40 to 0.54]
  Orthopnea - TFI | 0.54 [0.46 to 0.62]
  Orthopnea - HR | 0.59 [0.51 to 0.67]
  Orthopnea - RR | 0.55 [0.47 to 0.64]
  Fatigue - TFI | 0.57 [0.50 to 0.63]
  Fatigue - HR | 0.55 [0.48 to 0.62]
  Fatigue - RR | 0.47 [0.40 to 0.54]

5. Secondary Outcome: Correlation Between μCor Measurements and Subject Reported Symptoms - Number of Mild/Severe Symptoms
Description: as for outcome 4
Time Frame: 3 months
Population: The results indicate the number of mild or severe symptom reports preceded by a valid device measure. Each of the 245 participants in the study could contribute data to either Arm/Group depending on the severity of their symptoms across the 3-month study duration.
Measure: Number; unit: Symptoms
Groups:
- µCor Wearers With Mild Symptoms: Subjects wearing the µCor device with Mild Symptoms
- uCor Wearers With Severe Symptoms: Subjects wearing the uCor device with Severe Symptoms
Arm/Group | µCor Wearers With Mild Symptoms | uCor Wearers With Severe Symptoms
Number analyzed (Participants) | 245 | 245
Symptoms
  Dyspnea - TFI | 147 | 124
  Dyspnea - HR | 135 | 117
  Dyspnea - RR | 136 | 124
  Orthopnea - TFI | 206 | 65
  Orthopnea - HR | 190 | 57
  Orthopnea - RR | 197 | 64
  Fatigue - TFI | 134 | 141
  Fatigue - HR | 120 | 126
  Fatigue - RR | 128 | 130

6. Secondary Outcome: Frequency of Subject Reported Symptoms
Description: During weekly phone calls and monthly office visits, subjects reported whether they experienced new arrhythmia and/or heart failure symptoms. Results indicate the number of times that subjects reported each of these two symptoms.
Time Frame: 3 months
Population: 228 subjects completed at least one weekly phone call or monthly office visit case report form in which they could self-report arrhythmia and heart failure symptoms
Measure: Count of Participants; unit: Participants
Arm/Group | µCor Wearers
Number analyzed (Participants) | 228
Participants
  Frequency of self-reported arrhythmia symptoms: 0 Arrhythmia symptoms | 123
  Frequency of self-reported arrhythmia symptoms: 1 Arrhythmia symptom | 52
  Frequency of self-reported arrhythmia symptoms: 2 Arrhythmia symptoms | 22
  Frequency of self-reported arrhythmia symptoms: 3 Arrhythmia symptoms | 17
  Frequency of self-reported arrhythmia symptoms: 4 Arrhythmia symptoms | 3
  Frequency of self-reported arrhythmia symptoms: 5 Arrhythmia symptoms | 8
  Frequency of self-reported arrhythmia symptoms: 6+ Arrhythmia symptoms | 3
  Frequency of self-reported heart failure symptoms: 0 Arrhythmia symptoms | 83
  Frequency of self-reported heart failure symptoms: 1 Arrhythmia symptom | 62
  Frequency of self-reported heart failure symptoms: 2 Arrhythmia symptoms | 30
  Frequency of self-reported heart failure symptoms: 3 Arrhythmia symptoms | 21
  Frequency of self-reported heart failure symptoms: 4 Arrhythmia symptoms | 9
  Frequency of self-reported heart failure symptoms: 5 Arrhythmia symptoms | 10
  Frequency of self-reported heart failure symptoms: 6+ Arrhythmia symptoms | 13

7. Secondary Outcome: Timing of Subject Reported Symptoms
Description: During weekly phone calls and monthly office visits, subjects reported whether they experienced new arrhythmia and/or heart failure symptoms. Results indicate the median number of weeks until a subject's first symptom report of each type.
Time Frame: 3 months
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Weeks
Groups:
- uCor Wearers: Subjects wearing the uCor device
Arm/Group | uCor Wearers
Number analyzed (Participants) | 228
Weeks
  Time from start of study until first arrhythmia symptom report (median, interquartile range) | 4 [2 to 6]
  Time from start of study until first heart failure symptom report (median, interquartile range) | 3 [2 to 5]

8. Secondary Outcome: Severity of Subject Reported Symptoms
Description: Each subject was expected to undergo an in-person office visit at the site on months 0, 1, 2, and 3 in which they reported the severity of their heart failure symptoms. Results indicate the number of subjects reporting each severity level of each symptom at each office visit.
Time Frame: 3 months
Population: 245 subjects were enrolled in the study. Each subject was expected to undergo an in-person office visit at the site on months 0, 1, 2, and 3 in which they self-reported heart failure symptoms. Note that this analysis includes the initial office visit (month 0).
Measure: Count of Participants; unit: Participants
Groups:
- µCor Wearers - Month 0: Subjects wearing the µCor device during Month 0
- uCor Wearers - Month 1: Subjects wearing uCor during Month 1
- uCor Wearers - Month 2: Subjects wearing the uCor during Month 2
- uCor Wearers - Month 3: Subjects wearing the uCor during Month 3
Arm/Group | µCor Wearers - Month 0 | uCor Wearers - Month 1 | uCor Wearers - Month 2 | uCor Wearers - Month 3
Number analyzed (Participants) | 245 | 245 | 245 | 245
Participants
  Severity of Dyspnea: Continuous | 21 | 16 | 8 | 7
  Severity of Dyspnea: Frequent | 132 | 61 | 53 | 43
  Severity of Dyspnea: Seldom | 53 | 55 | 40 | 35
  Severity of Dyspnea: None | 31 | 31 | 28 | 26
  Severity of Dyspnea: No data | 8 | 82 | 116 | 134
  Severity of Orthopnea: Continuous | 21 | 15 | 8 | 6
  Severity of Orthopnea: Frequent | 72 | 35 | 16 | 18
  Severity of Orthopnea: Seldom | 62 | 44 | 40 | 24
  Severity of Orthopnea: None | 82 | 69 | 66 | 63
  Severity of Orthopnea: No data | 8 | 82 | 115 | 134
  Severity of Fatigue: Continuous | 35 | 22 | 19 | 16
  Severity of Fatigue: Frequent | 114 | 62 | 48 | 37
  Severity of Fatigue: Seldom | 55 | 50 | 41 | 37
  Severity of Fatigue: None | 33 | 29 | 22 | 21
  Severity of Fatigue: No data | 8 | 82 | 115 | 134

9. Secondary Outcome: Hospital Readmission Rate During the Study Period
Description: During weekly phone calls and monthly office visits, subjects reported whether they experienced a new hospitalization since their last call/visit. An adjudication committee of physicians determined whether each hospitalization was due to HF or not.
Time Frame: 3 months
Population: Number of subjects hospitalized primarily for heart failure within 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | µCor Wearers
Number analyzed (Participants) | 245
Participants | 50

10. Secondary Outcome: Hospital Readmission Rate During Previous 90 Days Prior to Enrollment in Study
Description: At the time of enrollment, subjects reported how many hospitalizations they experienced in the 90 days prior to enrollment. Results indicate the number of subjects who reported a hospitalization in this time window.
Time Frame: 3 months
Population: Number of subjects with a hospitalization in the 90 days prior to enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | µCor Wearers
Number analyzed (Participants) | 245
Participants | 206

11. Secondary Outcome: Hospital Readmission Rate During Previous 90 Days Prior to Enrollment in Study
Description: At the time of enrollment, subjects reported how many hospitalizations they experienced in the 90 days prior to enrollment. Results indicate the median number of hospitalizations reported per subject in this time window.
Time Frame: 3 months
Population: Number of hospitalizations per subject during the 90 days prior to enrollment
Measure: Median (Inter-Quartile Range); unit: Hospitalizations
Arm/Group | µCor Wearers
Number analyzed (Participants) | 245
Hospitalizations | 2 [1 to 2]

12. Secondary Outcome: Mortality, Heart Failure Related Events, and Health Care Utilization Data at Six Months and One Year Post Enrollment
Description: During weekly phone calls, monthly office visits, the 6-month phone call, and the 1-year phone call, subjects reported whether they experienced a hospitalization, ER visit, or unplanned doctor's office visit since the last call/visit. An adjudication committee of physicians determined whether each hospitalization was due to HF or not. On each subject's final date of study participation, their survival status was recorded.
Time Frame: 6 months and 1 year
Population: Subjects enrolled in the study at 6 months and 1 year
Measure: Number; unit: Participants
Groups:
- Subjects at 6 Months: Subjects at 6 months
- Subjects at 1 Year: Subjects at 1 year
Arm/Group | Subjects at 6 Months | Subjects at 1 Year
Number analyzed (Participants) | 245 | 245
Participants
  Mortality: Number of subjects reported dead | 21 | 31
  Heart Failure (HF) Related Events: Number of subjects with a hospital readmission for HF | 68 | 77
  Health Care Utilization: Number of subjects with a hospitalization for any reason | 127 | 137
  Health Care Utilization: Number of subjects with an Emergency Room visit for any reason | 109 | 117
  Health Care Utilization: Number of subjects with an unplanned doctor's office visit for any reason | 54 | 62

ADVERSE EVENTS:
Time Frame: 1 Year
Description: All adverse events in the study that were causally related to the use of μCor were recorded as adverse device effects (ADEs). Each ADE was classified by the investigator as anticipated or unanticipated and then assessed for seriousness. An unanticipated ADE was defined as any ADE not identified by nature, severity, or frequency prior to the study.
Arm/Group | µCor Wearers
All-Cause Mortality (participants affected / at risk) | 35/257
Serious Adverse Events (participants affected / at risk) | 1/257
Other Adverse Events (participants affected / at risk) | 149/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | µCor Wearers (N=257)
Procedural Complication to ECHO (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | µCor Wearers (N=257)
Discomfort (Product Issues) | 3 (3)
Skin Irritation (Skin and subcutaneous tissue disorders) | 146 (146)

LIMITATIONS AND CAVEATS:
This study was conducted from 8/17/2018 to 12/1/2022 and partially overlapped with the COVID-19 Pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT03476187/Prot_SAP_000.pdf